CLINICAL TRIAL: NCT01404962
Title: A Post Marketing Surveillance Study to Monitor the Reactogenicity and Safety of Vaxem™Hib When Administered According to the Prescribing Information in Korea
Brief Title: Safety of Haemophilus Influenza Type b Vaccine When Administered to Korean Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V37_11
Record Dates: First submitted 2011-07-25; First posted 2011-07-28 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2012-09

CONDITIONS: Haemophilus Influenzae Type B Infection
Keywords: Haemophilus influenza type b; children; Korea; vaccine; Prevention of haemophilus influenza type b
MeSH Terms: conditions — Haemophilus Infections

ARMS (1):
- Group 1 (Other)
  Interventions: Biological: Haemophilus influenza type b conjugate vaccine

INTERVENTIONS:
Biological: Haemophilus influenza type b conjugate vaccine — Primary series is 3 doses given to infants beginning at 2 months of age with an interval of 2 months apart (i.e. 2, 4 and 6 months of age). Booster vaccination consists of 1 dose and is given to toddlers 16 to 20 months of age. In this study, subjects will receive vaccination from routine primary care.

SUMMARY:
This is a multicenter, post marketing surveillance study which aims to evaluate the safety profile of haemophilus influenza type b vaccine when administered to Korean children according to the product insert.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children 2 months to 5 years of age scheduled to receive vaccination

Exclusion Criteria:

* Contraindications to Vaxem™Hib Korean Prescribing information

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 764 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events 28 days following vaccination | 29 days to 5 months

CONTACTS AND LOCATIONS:
Locations (5):
- South Korea (5):
  - Moon's Pediatrics Clinic, Gyeonggi-do
  - Wooriai Pediatrics clinic, Incheon
  - KyungHee University Hospital, Seoul
  - Hanil General Hospital, Seoul
  - Yonsei Pediatrics Clinic, Seoul